CLINICAL TRIAL: NCT05869006
Title: The Effect of Designed SIA Instrument Supported Interpersonal Relations-Based Group Practice on Psychological Well-Being and Creativity: A Randomized, Single-Blind, Placebo-Controlled Study
Brief Title: The Effect of Designed SIA Instrument Supported Interpersonal Relations-Based Group Practice on Psychological Well-Being and Creativity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Derya Küliğ Atabey, PhD, Ege University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: EGE-ATABEY-001
Record Dates: First submitted 2023-05-04; First posted 2023-05-22 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Psychological Stress; Psychology, Positive; Psychological Well-Being
Keywords: interpersonal relations theory; psychological well-being; psychiatric nursing; creativity
MeSH Terms: conditions — Stress, Psychological; Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: In a single-blind randomized controlled study, 3X4 split-plot design was used. A stratified randomization was carried out according to gender with 30 students who met the criteria for inclusion in the sample from the determined target group. The research was conducted with a total of 30 students, 10 of whom were in the intervention group, 10 in the placebo control group, and 10 in the control group. In order to evaluate the data, Psychological Well-Being Scale (PWS) and Creativity Scale (CS) were applied at time series points (pretest, posttest, 1st month follow-up and 3rd month follow-up).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): No attempt was made. Measurement tools were applied simultaneously with the placebo control group and intervention group before, after and during the follow-up.
  * pretest
  * final test
  * Evaluated by follow-up measurements.
- Placebo Control Group (Placebo Comparator): A symbolic intervention consisting of six sessions, which was different from the content of the sessions applied to the intervention group, did not have any curative and active content, and was carried out simultaneously with the intervention group as the application time, was applied.
  Sessions lasted approximately one hour. It was carried out once a week. It was completed in six weeks. In the sessions, the problems faced by nursing students due to distance education during the Covid-19 pandemic, professional difficulties, experiences, and issues related to their professional goals were discussed.
  The effectiveness of the semi-structured sessions;
  * pretest
  * symbolic group work
  * final test
  * evaluated by follow-up measurements.
  Interventions: Behavioral: Placebo group practice
- Intervention Group (Experimental): A semi-structured group study consisting of six sessions based on interpersonal relations supported by the designed SIA instrument was applied. Sessions lasted approximately one hour. One session per week was administered. It was completed in six weeks. The initiatives applied in the sessions were implemented based on Peplau's theory of Interpersonal Relations. Group work was supported by the SIA instrument and music therapy techniques were used. In addition, positive psychology and psychological well-being literature were examined in the creation of initiatives. The effectiveness of semi-structured sessions;
  * pretest
  * group interaction study consisting of six sessions
  * final test
  * evaluated by follow-up measurements.
  Interventions: Behavioral: Designed SIA Instrument Supported Interpersonal Relations-Based Group Practice

INTERVENTIONS:
Behavioral: Designed SIA Instrument Supported Interpersonal Relations-Based Group Practice — Group Practice
  Arms: Intervention Group
Behavioral: Placebo group practice — The placebo control group application was carried out simultaneously with the intervention group application, and the group application without active curative content was applied.
  Arms: Placebo Control Group

SUMMARY:
The goal of this interventional study is to examine the effect of group practice based on interpersonal relations supported by the designed SIA instrument on psychological well-being and creativity.The main questions it aims to answer are:

* Is group practice based on interpersonal relations supported by the designed SIA instrument effective in increasing the psychological well-being levels of individuals?
* Is group practice based on interpersonal relations supported by the designed SIA instrument effective in increasing the creativity levels of individuals? Group study consisting of 6 sessions was applied to the participants. Sessions were administered once a week. It took six weeks. The effect of group practice based on interpersonal relations, supported by the designed SIA instrument, on individuals' psychological well-being and creativity levels was investigated.

DETAILED DESCRIPTION:
This research was carried out to examine the effect of group practice based on interpersonal relations supported by the designed SIA instrument on psychological well-being and creativity.

In a single-blind randomized controlled trial, a 3x4 split-plot design was used. The sample group was determined in two stages. The target group consisted of those who had scores lower than the mean scores of the Psychological Well-Being Scale (PWS) total score obtained from the nursing students who accepted to participate in the study. A stratified randomization was carried out according to gender with 30 students who met the criteria for inclusion in the sample from the determined target group. The study was conducted with a total of 30 students, 10 of whom were in the intervention group, 10 in the placebo control group, and 10 in the control group. Research data were collected with Descriptive Information Form, Psychological Well-Being Scale (PWS) and Creativity Scale (CS). A group application based on Peplau's Interpersonal Relations Theory, supported by the SIA instrument, was applied to the individuals in the intervention group. It is a rhythm instrument with a water effect sound, designed by SIA researchers and has a national utility model registration certificate. Music therapy techniques were also used in practice. The application was completed in a total of six weeks, one session per week. The placebo control group application was carried out simultaneously with the intervention group application, and the group application without active curative content was applied. No intervention was applied to the control group. In order to evaluate the data, PWS and SR were applied at time series points (pretest, posttest, 1st month follow-up and 3rd month follow-up).

In the analysis of the data, Descriptive statistics, Normal distribution of the data related to continuous variables were evaluated with the Shapiro Wilk test of normality. One-way analysis of variance (ANOVA) or Kruskal-Wallis H test was used to compare the variances of more than two independent groups when the assumption of normality of continuous variables was met. Repeated measures ANOVA (repeated measure ANOVA) was used when the assumption of normality was provided in the in-group and between-group comparisons for repeated measures. In the absence of normality, the nonparametric test (Nonparametric Tests for the F1-LD-F1 Design) was used for repeated measurements. In cases where the group*time interaction was significant, evaluations independent of the time effect were made and repeated measures ANOVA and Friedman tests were used. A value of p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old,
* Agreeing to participate in the research and volunteering to go to the rhythm guitar featured group practice.
* Being in the second or third grade.
* To have a lower score than the PWS total score limits (X=356.52) obtained from all students in the sample pool.

Exclusion Criteria:

* Presence of obstruction in the sense organs

  * Having a self-reported mental illness diagnosis
  * Individuals included in the initiative group do not attend two or more sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2023-03-17 (Actual)

PRIMARY OUTCOMES:
"Psychological Well-Being Scale" scores | A total of five months of designed SIA instrument supported interpersonal relations-based group practice for intervention group
  Decreased "Psychological Well-Being Scale" scores of intervention group in post test and follow-up measurements after SİA instrument supported interpersonal relations-based group practice
"Creative Scale" scores | A total of five months of designed SIA instrument supported interpersonal relations-based group practice for intervention group
  Decreased "Creative Scale" scores of intervention group in post test and follow-up measurements after SİA instrument supported interpersonal relations-based group practice

CONTACTS AND LOCATIONS:
Overall Officials: Ayşegül DÖNMEZ, Prof. Dr., Study Director — Ege University Faculty of Nursing; Derya KÜLİĞ ATABEY, PhD, Principal Investigator — Ege University Hospital (Application and Research Center)
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No